CLINICAL TRIAL: NCT06738888
Title: Renovated Prediction Model for Difficult. Transoral and Submental Endoscopic Thyroidectomy
Brief Title: Renovated Prediction Model for Difficult Transoral and Submental Endoscopic Thyroidectomy
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Ling Zhan, Principal Investigator, Shanghai 6th People's Hospital
Other Study IDs: 2025-KY-029(K)
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Cancer; Thyroid Diseases; Thyroid Nodule
Keywords: Endoscopic thyroidectomy; Transoral and submental approach; Prediction model
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases; Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Difficult transoral and submental thyroidectomy: (1) operative time more than 75% of the overall study cases (2) severe intraoperative injuries :: vascular injury, recurrent laryngeal nerve injury, trachea injury, esophagus injury
  Interventions: Other: Observations on clinicopathological factors influencing the difficulty of surgery
- Normal transoral and submental thyroidectomy: the remaining of the entire study cases excluding the difficult cases
  Interventions: Other: Observations on clinicopathological factors influencing the difficulty of surgery

INTERVENTIONS:
Other: Observations on clinicopathological factors influencing the difficulty of surgery — Age, body mass index, gender, thyroid function parameters, lesion size, lesion location, ultrasound data, thyromental distance, neck circumference, sternomental distance, ratio of height-to-thyromental distance, RHTMD, ratio of height-to-sternomental distance, RHSMD

SUMMARY:
The investigators have previously proposed a prediction model for difficult transoral and submental thyroidectomy through a retrospective study. In order to better promote transoral and submental endoscopic approach for thyroid surgery and to set up an appropriate training course, the investigators aim to renovate and validate the prediction model through a prospective study.

DETAILED DESCRIPTION:
Male sex, age, BMI, neck length and certain thyroid disease such as thyroiditis and hyperthyroidism have been long cited as indicators of a difficult thyroidectomy. The investiagtors hypothesized that neck extension was critical to the exposure and visualization of the surgical field in the endoscopic thyroidectomy. Therefore, several measurements were innovatedly integrated into the prediction model, including neck circumference, thyromental distance, sternomental distance, ratio of height-to-thyromental distance, ratio of height-to-sternomental distance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of differentiated thyroid cancer with a maximum diameter not exceeding 4 cm
* Clinical diagnosis of benign thyroid nodule with a maximum diameter not exceeding 6 cm
* Absence of suspicious lateral lymph nodes or distant metastases

Exclusion Criteria:

* Participants with fusion or fixation of lymph nodes in the neck
* Participants with history of neck surgery or radiation
* Participants with vocal fold fixation by preoperative fibrolaryngoscope
* Participants with preoperative examination suggestive of extrathyroidal invasion
* Participants with a significantly restricted neck and/or jaw

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with FNA proven differentiated thyroid cancer, were willing to undergo thyroidectomy and central lymph node dissection via transoral and submental approach. Patients were well informed about the transoral and submental approach and were aware of the potential benefits and risks. Patient consented for us to use perioperative data.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
1.Number of participants with recurrent laryngeal nerve injury 1.Number of participants with recurrent laryngeal nerve injury Number of participants with recurrent laryngeal nerve injury | through study completion, an average of 1 year
  impaired vocal cord mobility confirmed by postoperative laryngoscopy
Number of participants with hypoparathyroidism Number of participants with hypoparathyroidism Number of participants with hypoparathyroidism | through study completion, an average of 1 year
  a postoperative parathyroid hormone level of less than 10 pg/ml
  a postoperative parathyroid hormone level of less than 10 pg/ml a postoperative parathyroid hormone level of less than 10 pg/ml
Number of participants with mental nerve injury | through study completion, an average of 1 year
  a postoperative numbness in the lower lip and submental area
operative time | immediately at the end of the surgery
  operative time was defined as the duration from incision to closure, and was collected from anesthesia record sheet

SECONDARY OUTCOMES:
hospitalization | Length of stay from hospitalisation to discharge
  days of hospitalization
degree of pain | approximately 4 hours after surgery and on postoperative day 1
  pain intensity was assessed using a standard visual analogue score, with a score of 0 to 10 corresponding to no pain to the most severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Ling Zhan, Doctor, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
Data are available on request due to privacy or other restrictions. The data that support the findings of this study are available on request from Ling Zhan. The data are not publicly available due to them containing information that could compromise research participant privacy.